CLINICAL TRIAL: NCT07271823
Title: Establishment of a Predictive Model for Immunotherapy Response in Pancreatic Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ying Jieer, Principal Investigator, Zhejiang Cancer Hospital
Other Study IDs: IRB-2024-974（IIT）
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer Non-resectable
Keywords: Chemotherapy combined with immunotherapy; Pancreatic Cancer Non-resectable; efficacy prediction; Biomarker
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Patient tumor tissue sections, plasma, serum, and stool specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Locally advanced or metastatic pancreatic ductal adenocarcinoma: Locally advanced or metastatic pancreatic ductal adenocarcinoma in patients who have not previously received systemic anticancer therapy
  Interventions: Other: Sample Collection

INTERVENTIONS:
Other: Sample Collection — Prior to treatment initiation (baseline), collect tissue specimens from the patient's pancreatic cancer or liver metastases via ultrasound-guided biopsy. Simultaneously collect one tube of EDTA-anticoagulated peripheral blood, one tube of clotting-anticoagulant peripheral blood, and one stool sample. Collect peripheral blood and stool samples at key time points including initial assessment, second assessment, and disease progression. Plasma and serum were extracted from the two tubes of peripheral blood. Concurrently, clinical and pathological parameters (age, sex, tumor TNM staging, pathological findings, etc.) and follow-up prognostic information (recurrence status, survival time) were recorded.

SUMMARY:
This project aims to establish a single-center, prospective, observational clinical cohort for pancreatic cancer immunotherapy. It plans to enroll 100 patients with advanced pancreatic cancer, collecting tumor tissue sections, plasma, serum, and fecal samples. Through multi-omics analysis including proteomics, metabolomics, and microbiomics, the project will develop predictive models for immunotherapy response.

DETAILED DESCRIPTION:
Primary Objective: Establish a cohort for immunotherapy combined with chemotherapy in advanced pancreatic cancer, ultimately developing predictive models for immunotherapy response based on proteomics, metabolomics, and microbiome data.

Secondary Objectives: Map the clinical and genomic/metabolomic/microbiome profiles of patients with advanced pancreatic ductal adenocarcinoma, evaluate the therapeutic efficacy of immunotherapy combined with chemotherapy, and explore potential biomarkers for predicting immunotherapy response.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Histologically or cytologically confirmed locally advanced or metastatic pancreatic ductal adenocarcinoma that is unresectable;
3. No prior systemic anticancer therapy;
4. At least one measurable lesion confirmed according to RECIST 1.1 criteria;
5. Receiving first-line treatment with an immunotherapy combined with chemotherapy regimen;
6. Signed informed consent.

Exclusion Criteria:

1. Active malignancy other than pancreatic cancer within the past 5 years or concurrently;
2. Prior receipt of immunotherapy or anti-angiogenic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced or metastatic pancreatic ductal adenocarcinoma confirmed histologically or cytologically as unresectable
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Best Tumor Response | 12 months
  Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria.
Overall Survival | 60 months
  Overall survival is the duration from diagnosis to death. For patients who are alive, overall survival is censored at the last contact.

SECONDARY OUTCOMES:
Progression-free Survival | 36 months
  The period from diagnosis until disease progression or death on study, whichever occurred first.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Zhejiang, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided
We currently have no plans to share individual participant data (IPD) with other researchers.